CLINICAL TRIAL: NCT07172867
Title: A Randomized, Double-Blind, Placebo-Controlled Multicenter Phase 2 Study to Evaluate the Safety, Efficacy and Tolerability of Ofirnoflast (HT-6184) and Semaglutide in Obese or Overweight Participants With Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Ph2 Study to Evaluate the Safety, Efficacy and Tolerability of HT-6184 and Semaglutide in Obese Participants With T2DM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Halia Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HT-6184-IIO-001
Record Dates: First submitted 2025-08-25; First posted 2025-09-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HT-6184 2mg Treatment (Experimental): Ofirnoflast (2 mg): dosed once a day, orally (PO QD) + semaglutide (1 mg): dosed weekly (q1wk), via subcutaneous (SC) injection for 12 weeks.
  Interventions: Drug: HT-6184; Drug: Semaglutide 1 mg
- HT-6184 2mg Matching Placebo (Placebo Comparator): Placebo: dosed once a day, orally (PO QD) + semaglutide (1 mg): dosed weekly (q1wk), via SC injection for 12 weeks.
  Interventions: Drug: HT-6184 Matching Placebo; Drug: Semaglutide 1 mg

INTERVENTIONS:
Drug: HT-6184 — 2mg QD
  Arms: HT-6184 2mg Treatment
Drug: HT-6184 Matching Placebo — 2mg QD
  Arms: HT-6184 2mg Matching Placebo
Drug: Semaglutide 1 mg — Semaglutide 1 mg, every week

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ofirnoflast in combination with semaglutide in comparison to semaglutide alone in obese participants with T2DM.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and safety of ofirnoflast in combination with semaglutide in comparison to semaglutide alone in obese participants with T2DM.

This study is a randomized, double-blind, placebo-controlled, parallel-group clinical trial.

* The study duration will be up to 28 weeks.
* The screening period will be up to 4 weeks
* The treatment duration will be 12 weeks.
* The follow-up period will be 12 weeks
* The visit frequency will be every 4 weeks during the treatment phase of the study.
* There will be an anticipated 7 scheduled clinic visits, including 1 screening visit and 2 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* BMI between 27 kg/m2 and 40 kg/m2.
* Stable body weight (± 5 kg) within 90 days of screening, and body weight <150 kg.
* HbA1c is 7.5-10.5% at screening.
* Established diagnosis of T2DM.
* Receiving a stable 1mg SC q1wk dose of semaglutide (Ozempic®) for ≥ 90 days prior to signing informed consent.
* Females must meet one of the following:

  1. Postmenopausal (>45 years of age with amenorrhea for at least 12 months, without using exogenous hormonal contraception and with FSH ≥ 40 IU/L).
  2. Surgically sterile (hysterectomy, bilateral salpingectomy; oophorectomy) for at least 6 months.
  3. Using a double contraception including a barrier method (condom, diaphragm, or occlusive cap) and a highly effective method of birth control, which includes the following:

  i. Established use (i.e. at least 90 days prior to signing of ICF) of combined (estrogen and progestogen) oral, intravaginal, or transdermal hormonal contraceptive associated with inhibition of ovulation ii. Established use (i.e. at least 90 days prior to signing of ICF) of progestogen-only oral, injectable, or implantable hormonal contraceptive associated with inhibition of ovulation iii. Established use (i.e. at least 90 days prior to signing of ICF) of an intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) iv. Bilateral tubal occlusion completed at least 90 days prior to signing of ICF d. Vasectomized partner with the appropriate post-vasectomy documentation of the absence of spermatozoa in the ejaculate. Participant must provide documentation before the first dose of ofirnoflast (study day 1).

  e. Sexual abstinence, when this is in line with the preferred and usual lifestyle of the participant
* Male participants who are sexually active with a woman of childbearing potential must agree to use a double contraception including a barrier method (male condom) and a highly effective method of contraception (highly effective methods of contraception are listed above) during the study and for 30 days after the last dose of ofirnoflast/ placebo.
* In the case of WOCBP, participants must have a negative serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at screening and negative urine pregnancy tests on first day of dosing and at each study visit.
* Able to comply with the study procedures in the view of the Investigator.

Exclusion Criteria:

* Any prescription or over-the-counter medications intended for weight loss within 6 months of screening, excluding semaglutide.
* History of, or known hypersensitivity to, monoclonal antibody drugs or a contraindication to semaglutide (e.g. Ozempic® or Wegovy®)
* Use of other investigational drugs at the time of screening or within 30 days or 5 half-lives prior to signing of the ICF, whichever is longer, or longer if required by local regulations
* Previous or current diagnosis of Type 1 diabetes mellitus (T1DM) or current gestational diabetes.
* Diagnosis of T2DM requiring current use of insulin, repaglinide, saxagliptin, and sulfonylureas.

Note. Use of Metformin for the purposes of glycemic control is not exclusionary.

* History of diabetic ketoacidosis (within 90 days of screening), or proliferative or severe retinopathy (i.e., retinopathy requiring acute treatment).
* Previous bariatric surgery, liposuction, or planned weight loss surgery.
* Current or past diagnosis of pancreatitis
* Current or past diagnosis of severe gastroparesis
* Personal or within first-degree relative family history of medullary thyroid cancer or multiple endocrine neoplasia type 2
* Calcitonin ≥20 ng/L measured by central laboratory at screening (individuals with elevated calcitonin at initial screening may be re-screened)
* Laboratory abnormalities at screening
* Current or history of clinically significant (per Investigator's judgment) liver or biliary disease or significantly abnormal LFT at screening (see above)
* Current acute or chronic self-reported HCV and/or HBV infection
* Current or history of clinically significant renal disease (per Investigator's judgment) or eGFR<60mL/min/1.73m2
* Prior history of malignancy (including breast cancer, lymphoma, leukemia) within the past 5 years except for cervical carcinoma in situ that has been completely resected with no evidence of recurrence or metastatic disease for at least 12 months or cured basal cell carcinoma with no evidence of recurrence for at least 12 months.
* History of a major organ transplant (e.g. kidney, heart, liver, lung) or hematopoietic stem cell/ bone marrow transplant.
* History of lymphoproliferative disease or signs/ symptoms suggestive of possible lymphoproliferative disease, including splenomegaly of lymphadenopathy.
* History or current moderate to severe congestive heart failure (New York Heart Association class III or IV), or within the last 6 months, a cerebrovascular accident, myocardial infarction, unstable angina, unstable arrhythmia or any other cardiovascular condition which, in the opinion of the Investigator, would put the participant at risk by participation in the study.
* Undergone any major surgery within 8 weeks prior to study entry or will require major surgery during the study that, in the opinion of the Investigator, would pose an unacceptable risk to the participant.
* Planning elective surgery during the study duration
* Inherited or acquired thrombophilia and/ or current or history of thromboembolic events/ disease.
* Screening 12-lead ECG that demonstrates relevant abnormalities that, in the opinion of the Investigator, are clinically significant and indicate an unacceptable risk for the participant's participation in the study (e.g., QTc >450 msec or a QRS interval >120 msec). If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the participant's eligibility.
* History or evidence of any other clinically significant concomitant disorder, condition or disease that, according to the Investigator's and medical monitor's (if consulted) judgment, would pose a risk to participant safety or interfere with the study evaluation, procedures, completion or interpretation of data
* Pregnant or breast-feeding.
* Blood donation within the last month before study day 1 (first dose of ofirnoflast or placebo)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assess glycemic control using HbA1c (%) | From first dose through End of Study (up to 12 weeks per participant)
  Evaluate glycemic control using HbA1c (%) from baseline to week 12 in participants treated with ofirnoflast or placebo in combination with semaglutide. This outcome will assess if the participant was able to reduce HbA1c by at least 1.5%.
Assess weight loss using body weight measurements | From first dose through End of Study (up to 12 weeks per participant)
  Evaluate weight loss using body weight measurements from baseline to week 12 in participants treated with ofirnoflast or placebo in combination with semaglutide. This outcome will assess if the participant was able to reduce body weight by at least 5%.

SECONDARY OUTCOMES:
Assess the change in HbA1c (% point) | From first dose through End of Study (up to 12 weeks per participant)
  Evaluate the change in HbA1c (% point) from baseline to week 12 in participants treated with ofirnoflast or placebo in combination with semaglutide.
Assess the change in body composition utilizing DEXA body scan | From first dose through End of Study (up to 12 weeks per participant)
  Evaluate the change in body composition utilizing DEXA body scan from baseline to week 12 in participants treated with ofirnoflast or placebo in combination with semaglutide.
Assess the PK profile; AUC 0-inf, AUC 0-last, AUC tau, Cmax, tmax, t1/2, and Cl/F | From first dose through End of Study (up to 12 weeks per participant)
  Evaluate the PK profile (AUC 0-inf, AUC 0-last, AUC tau, Cmax, tmax, t1/2, and Cl/F) of ofirnoflast in participants treated with ofirnoflast and semaglutide
Assess number of participants who experience Serious Adverse Events (SAEs) | From first dose through End of Study (up to 12 weeks per participant)
  The safety and tolerability of ofirnoflast or placebo in combination with semaglutide will be evaluated based on the incidence of SAE in participants, as assessed according to CTCAE v5.0. The number of participants who experience a SAE will be reported.
Assess number of participants who experience treatment emergent adverse events (TEAEs) | From first dose through End of Study (up to 12 weeks per participant)
  The safety and tolerability of ofirnoflast or placebo in combination with semaglutide will be evaluated based on the incidence of TEAE in participants, as assessed according to CTCAE v5.0. The number of participants who experience a TEAEs will be reported.
Assess number of participants who experience treatment related adverse events (TRAEs) | From first dose through End of Study (up to 12 weeks per participant)
  The safety and tolerability of ofirnoflast or placebo in combination with semaglutide will be evaluated based on the incidence of TRAEs in participants, as assessed according to CTCAE v5.0. The number of participants who experience a TRAEs will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No